CLINICAL TRIAL: NCT03694730
Title: Continued Activity During Rehabilitation in Patients With Patellar Tendinopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Delaware (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1217479
Record Dates: First submitted 2018-10-01; First posted 2018-10-03 (Actual); Last update posted 2021-03-09 (Actual); Status verified 2021-03

CONDITIONS: Patellar Tendinopathy; Patellar Tendinitis; Patellar Tendon Pain; Patellar Tendinosis; Jumper's Knee
Keywords: Tendinopathy; Tendinitis; Tendinosis; Rehabilitation; Exercise Treatment; Activity Modification
MeSH Terms: conditions — Tendinopathy | interventions — Exercise Therapy; Physical Therapy Modalities

STUDY DESIGN:
Intervention Model Description: Two treatment groups receiving different activity modification instructions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pain-guided Activity Modification (Experimental): Participants in the Pain guided Activity Modification group will receive an exercise program consisting of progressive patellar tendon loading exercises Outside of physical therapy treatment, these participants will modify activity based on the Pain-Monitoring Model.
  Interventions: Other: Exercise Treatment; Other: Pain- Guided Activity Modification
- Pain-free Activity Modification (Active Comparator): Participants in the Pain-free Activity Modification group will receive an identical exercise program to the Pain-guided Activity Modification group. However, participants will not be allowed to participate in activities that cause patellar tendon pain or excessively load the patellar tendon (e.g. jumping) outside of physical therapy treatment.
  Interventions: Other: Exercise Treatment

INTERVENTIONS:
Other: Exercise Treatment — Exercise treatment will consist of squatting and knee extension exercises, designed to progressively load the patellar tendon (Heavy-Slow Resistance protocol). A pain-monitoring model is used to guide exercise loads. As the protocol progresses, exercise load is increased while repetitions are decreased.
  Other Names: Rehabilitation exercise; Physical Therapy treatment
Other: Pain- Guided Activity Modification — Participants sports participation and physical activity will be guided by the Pain-Monitoring Model. Using the Pain-Monitoring Model, patients may participate in activities that cause patellar tendon pain, as long as pain does not exceed 5/10 on the numeric pain rating scale (NPRS) (0 = No pain, 10 = Worst pain imaginable) during or immediately after activity. Additionally, pain should return to pre-activity levels by the following morning and pain should not increase from week-to-week.
  Arms: Pain-guided Activity Modification

SUMMARY:
This pilot study will evaluate the feasibility of pain-guided activity modification during rehabilitation for patellar tendinopathy. The information provided will be utilized to conduct a larger randomized clinical trial to determine if there is a difference in recovery from patellar tendinopathy during rehabilitation between individuals that use pain-guided activity modification and those that halt all painful activities. Recovery from patellar tendinopathy will be assessed using pain ratings, tendon-specific outcome measures, tendon structure, tendon mechanical properties, and muscle function.

DETAILED DESCRIPTION:
Patellar tendinopathy is a chronic, degenerative condition of the patellar tendon that results in pain, altered tendon structure, functional impairments, decreased sports performance, and lost playing time. It commonly affects jumping athletes in sports such as volleyball and basketball. The prevalence of patellar tendinopathy is high, with 11.8-14.4% of recreational and 32-45% of elite volleyball and basketball players reporting symptoms. Although many athletes will seek treatment, 27-49% will experience re-injury and over half of those injured will retire from their sport of choice due to recurrent symptoms. Additionally, the absence of symptoms does not ensure full recovery of tendon health and function, which may contribute to the high rates of recurrence.

Exercise therapy for the treatment of patellar tendinopathy is supported by the highest level of evidence. However, exercise therapy has been found to be ineffective if the patients continue with full sports participation. On the other hand, it is unclear if it is necessary for athletes to completely halt physical activities while undergoing treatment. Absence from sport due to injury has been associated with increased anxiety, depression, and decreased self-esteem. Therefore, it is of interest to maintain sports participation, as long as it does not interfere with injury recovery.

In a randomized controlled trial (RCT) the investigators evaluated if continued running and jumping during treatment with an Achilles tendon-loading strengthening program had an effect on the outcome in patients with Achilles tendinopathy. In this study the investigators found that there were no detrimental effects of being physically active when the level of activity was guided by a pain-monitoring model. However, the impact of pain-guided activity modification has not been investigated in patellar tendinopathy. The proposed pilot study will determine if continued activity, using a pain-monitoring model, is feasible during treatment for patients with patellar tendinopathy. Furthermore, the investigators will evaluate if there is a negative effect on recovery of symptoms, tendon structure and mechanical properties, and functional recovery when adding continued physical activity compared to rest during exercise therapy treatment. To achieve this objective, the investigators will conduct a RCT comparing patients with patellar tendinopathy that are allowed to continue sports participation during treatment, using a pain-monitoring model, to those that are not allowed to participate in activities that cause pain.

Aim 1 is to evaluate feasibility by examining compliance and satisfaction with continued sports participation, guided by a pain-monitoring model, compared to refraining from sports participation during treatment. This will provide critical information to determine if a larger randomized clinical trial is feasible and if the study protocol needs to be modified. Aim 2 is to evaluate if there is a difference in change over time in symptoms, tendon structure and mechanical properties, and function between the two interventions.

This study will be the first to evaluate continued sports participation, guided by a pain-monitoring model, during rehabilitation in patients with patellar tendinopathy. The results from this study will play a critical role in achieving the long-term research goal of understanding of how to develop tailored treatments for patients with tendon injury. Ultimately this work will inform clinician recommendations regarding activity modification and potentially, limit the negative psychosocial impacts of the injury.

ELIGIBILITY:
Inclusion Criteria:

* Physically active individuals with a diagnosis of patellar tendinopathy

Exclusion Criteria:

* Injury that limits ability to participate in testing
* History of knee surgery within the last 6 months.
* Injection, shockwave, tenotomy or Ten-X to the patellar tendon within the last 6 months.

Ages: 16 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Actual)
Dates: Start 2018-03-11 (Actual); Primary Completion 2020-04-15 (Actual); Study Completion 2020-04-15 (Actual)

PRIMARY OUTCOMES:
Willingness to Participate | Percentage over initial year of study recruitment
  The percentage of potential participants that are willing to enroll and be randomized to one of the two groups after being informed of the study
Drop Out Rate | Percentage over initial year of study recruitment
  The percentage of participants that drop-out after study randomization.
Symptoms | Change over time with evaluations at baseline, 6-weeks, and 12-weeks
  Victorian Institute of Sport Assessment - Patella questionnaire (VISA-P)
Tendon Structure | Change over time with evaluations at baseline, 6-weeks, and 12-weeks
  Ultrasound imaging of tendon structure
Continuous Shear Wave Elastography (cSWE) to measure tendon mechanical properties | Change over time with evaluations at baseline, 6-weeks, and 12-weeks
  Continuous shear wave elastography (cSWE) will be used to measure shear modulus, viscosity and dynamic shear modulus of the patellar tendon.
Muscle-tendon function | Change over time with evaluations at baseline, 6-weeks, and 12-weeks
  Functional test battery consisting of two jump tests, one muscle strength and activation test.

SECONDARY OUTCOMES:
Adverse Events | Number over first year of study recruitment
  The number and types of adverse events occurring in either group during study participation.
Knee Injury and Osteoarthritis Outcome Score - Quality of Life subscale (KOOS-QOL) | Change over time with evaluations at baseline, 6-weeks, and 12-weeks
  The Knee Injury and Osteoarthritis Outcome Score - Quality of Life subscale (KOOS-QOL) will be used to assess the impact of knee injury on quality of life. The KOOS-QOL is a subscale of the Knee Injury and Osteoarthritis Outcome Score (KOOS). Scores range from 0 to 100 with 0 indicating extreme detrimental effect on quality of life and 100 indicating no effect on quality of life.
Tampa Scale of Kinesiophobia (TSK) | Change over time with evaluations at baseline, 6-weeks, and 12-weeks
  The Tampa Scale of Kinesiophobia (TSK) will be used to measure participants fear of movement and re-injury (kinesiophobia). Scores on the TSK range from 17 to 68 with 17 indicating minimal to no fear of movement and re-injury and 68 indicating very high fear of movement and re-injury.
Pain Catastrophizing Scale (PCS) | Change over time with evaluations at baseline, 6-weeks, and 12-weeks
  The Pain Catastrophizing Scale (PCS) will be used to assess patients pain catastrophizing. Scores on the PCS range from 0 to 52 with 0 indicating no pain catastrophizing and 52 indicating high levels of pain catastrophizing.
Numeric Pain Rating Scale (NPRS) | Change over time with evaluations at baseline, 6-weeks, and 12-weeks
  Patellar tendon pain will be assessed using the numeric pain rating scale. Participants are asked to verbally rate their pain on a scale of 0 to 10 with 0 indicating "No pain at all" and 10 indicating the "Worst pain imaginable".
Depression, Anxiety and Stress Scale (DASS-21) | Change over time with evaluations at baseline, 6-weeks, and 12-weeks
  Participant's depression, anxiety and stress levels will be assessed using the Depression, Anxiety and Stress Scale (DASS-21). The DASS-21 consists of three subscales, (1) Depression, (2) Anxiety, and (3) Stress. Scores for each subscale range form 0 to 42, where 0 indicates normal levels of the measured trait (depression, anxiety or stress) and 42 indicates extremely severe levels of the measured trait.
Compliance with Activity Modification | Average compliance rate for each group over first year of study recruitment
  Training log - Number of times pain exceeded pain threshold for either group

CONTACTS AND LOCATIONS:
Locations (1):
- University of Delaware, Newark, Delaware, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sprague AL, Couppe C, Pohlig RT, Snyder-Mackler L, Silbernagel KG. Pain-guided activity modification during treatment for patellar tendinopathy: a feasibility and pilot randomized clinical trial. Pilot Feasibility Stud. 2021 Feb 25;7(1):58. doi: 10.1186/s40814-021-00792-5. PMID 33632313
- See also: Delaware Tendon Research Group — https://sites.udel.edu/pt/research/karin-gravare-silbernagel-pt-phd-atc/